CLINICAL TRIAL: NCT00749099
Title: 092206: Bioavailability of Pancreatic Enzymes in the Human Upper Intestine (Duodenum and Jejunum) From PANCRECARB® (Pancrelipase), Delayed Release Capsules, Buffered and Enteric-Coated Microspheres
Brief Title: Bioavailability of Pancreatic Enzymes in the Human Upper Intestine (Duodenum and Jejunum)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: No longer required study by FDA for NDA approval.
Sponsor: Digestive Care, Inc. (Industry)
Collaborators: St. Louis University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: DCI092206; IRB #14687
Record Dates: First submitted 2008-09-07; First posted 2008-09-09 (Estimated); Last update posted 2013-02-22 (Estimated); Status verified 2013-02

CONDITIONS: Exocrine Pancreatic Insufficiency
MeSH Terms: conditions — Exocrine Pancreatic Insufficiency | interventions — Pancrelipase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Phase I (Placebo Comparator): All subject participate in Phase I
  Interventions: Drug: placebo
- Phase II (Active Comparator): All subject participate in Phase II
  Interventions: Drug: pancrelipase

INTERVENTIONS:
Drug: pancrelipase — The test drug (PANCRECARB® [pancrelipase] - Phase II) with a standardized Lundh meal.
  Gastric samples are collect once an hour and duodenal samples are collected every 15 minutes for each phase (4 hours each).
  Other Names: PANCRECARB®
  Arms: Phase II
Drug: placebo — 5 capsules of a placebo drug (Phase I) with a standardized Lundh meal.
  Gastric samples are collect once an hour and duodenal samples are collected every 15 minutes for each phase (4 hours each).
  Arms: Phase I

SUMMARY:
The overall purpose of this research is to demonstrate (or measure) the intestinal availability of lipase, amylase, and protease (enzymes the body has a shortage of) from PANCRECARB® when administered with a meal.

DETAILED DESCRIPTION:
Eligible patients for this placebo-controlled study had confirmed exocrine pancreatic insufficiency with a stool pancreatic elastase of <75 mcg/g. Patients who satisfied all inclusion criteria are prepared for endoscopic placement of three Liguory nasal biliary aspiration catheters: one 8.5 fr. catheter in the distal duodenum for aspiration, one 7.0 fr. catheter in the first portion of the duodenum for infusion of a PEG marker (4 mL/min) and one 7.0 fr. in the stomach for aspiration. Baseline samples are obtained from the gastric and distal duodenal ports and placed on ice. Subjects are then asked to swallow 5 capsules of a placebo (Phase I) or the test drug (PANCRECARB® (pancrelipase) - Phase II) with a standardized Lundh meal. Gastric samples are collected once an hour and duodenal samples are collected every 15 minutes for each phase (4 hours each). All collected samples were tested for the following parameters to demonstrate bioavailability of enzymes originating from PANCRECARB® (pancrelipase): lipase, amylase and protease activities, pH (bicarbonate), and protein fingerprinting by SDS-PAGE analysis.

ELIGIBILITY:
Inclusion Criteria:

* Documented chronic pancreatitis, alcohol induced chronic pancreatitis or cystic fibrosis
* Documented pancreatic enzyme insufficiency as determined by spot fecal elastase-1 <75 mcg/g stool at the time of inclusion in the study
* Required daily exogenous enzyme supplementation with commercially available pancreatic enzymes
* > 18 years of age
* Male and female subjects qualify
* Able to swallow capsules
* Clinically stable with no evidence of an acute medical condition
* History of steatorrhea

Exclusion Criteria:

* History of fibrosing colonopathy in CF subjects
* Current diagnosis or a history of distal intestinal obstruction syndrome (DIOS) in the past 4 months
* Known contraindication, sensitivity or hypersensitivity to porcine pancreatic enzymes
* Active liver disease
* ALT or AST >3 times the upper limit of normal
* Bilirubin >3 times the upper limit of normal
* Acute pancreatitis or acute exacerbation of chronic pancreatitis
* Acute treatment with any systemic (oral or IV) antibiotics two weeks prior to screening
* Subjects on erythromycin unwilling to discontinue the treatment two weeks prior to screening
* Receiving treatment with antacids or H2 receptor blockers or proton pump inhibitors and unable to discontinue these treatments prior to day 1
* Inability to cooperate with or non-compliant with required study procedures
* Pregnant, breast feeding
* Current daily prescribed scheduled use of narcotics (patients requiring PRN use of narcotics are not excluded)
* Poorly controlled diabetes
* A medical condition which the investigator deems significant enough to interfere with the ability of the subject to participate in the intubation study or interfering with assessment or enzyme bioavailability
* Stomach pH > 4
* Small bowel disease (i.e. celiac disease)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2007-04; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Evidence of the bioavailability of lipase, amylase and protease in the upper intestine from exogenously administered PANCRECARB® (pancrelipase), when taken with a Lundh test meal. | 4 hours post administration of PANCRECARB® and or Placebo